CLINICAL TRIAL: NCT01311960
Title: Topical Bevacizumab 0.05% Eye Drops for Preventing Recurrent Pterygium, A Randomized, Double-masked, Controlled Trial
Brief Title: Topical Bevacizumab for Preventing Recurrent Pterygium
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Chulalongkorn University (Other)
Responsible Party: Principal Investigator, Ngamjit Kasetsuwan, Associated professor, Chulalongkorn University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: IRB No. 227/53
Record Dates: First submitted 2010-12-01; First posted 2011-03-10 (Estimated); Last update posted 2013-04-09 (Estimated); Status verified 2011-03

CONDITIONS: Pterygium; Bevacizumab; VEGF; Anti-VEGF
Keywords: pterygium; recurrent pterygium; bevacizumab; VEGF; anti-VEGF
MeSH Terms: conditions — Pterygium | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- bevacizumab eye drop (Experimental)
  Interventions: Drug: bevacizumab eye drop 0.05%
- placebo normal saline eye drop (Experimental)
  Interventions: Drug: normal saline 0.9%

INTERVENTIONS:
Drug: bevacizumab eye drop 0.05% — bevacizumab eye drop 0.05% will apply 4 times a day for 3 months
  Other Names: Study arm
  Arms: bevacizumab eye drop
Drug: normal saline 0.9% — normal saline eye drop 0.9% will apply 4 times a day for 3 months.
  Other Names: placebo arm
  Arms: placebo normal saline eye drop

SUMMARY:
The purpose of this study is to determine whether bevacizumab eye drop is effective in the treatment of recurrent pterygium.

DETAILED DESCRIPTION:
A pterygium is a degenerative and proliferative fibrovascular disorder of the ocular surface. Patients may be asymptomatic, irritation, decreased vision, diplopia or limit ocular movement. The mainstay treatment is surgical removal of the head, neck and body of the pterygium. However, if there is no adjunctive treatment, the recurrence is unacceptably high which is 63% in general. Various adjunctive measures are applied to prevent recurrence including use of mitomycin C, beta-irradiation and surgical methods such as conjunctival and amniotic membrane graft. However, each method has its advantages and disadvantages.

The histologic finding of recurrent pterygium often has aggressive fibrovascular growth. Vascular endothelial growth factor(VEGF)has been detected in increased amounts in pterygium tissue, compared with normal conjunctiva and it is also correlated with post-operative recurrence. Bevacizumab, an Anti-VEGF, binds to VEGF and prevents the interaction of VEGF to its receptors on the surface of vascular endothelial cells. Administration of bevacizumab leads to inhibition of endothelial cell proliferation and new blood vessel formation. Even though there are reported the efficacy of topical bevacizumab in inhibiting the impending recurrent pterygium, there is no study for preventing recurrence after primary pterygium removal.

We conduct a prospective, randomized, double-masked, controlled trial to evaluate the efficacy of topical bevacizumab 0.05% eye drops for preventing recurrence in primary pterygium.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are diagnosed with primary pterygium and plan for pterygium excision with bare sclera by single surgeon. (G.N.)
* Patients with pterygium who understand and can follow the study protocol.
* Patients of age more than 30 years

Exclusion Criteria:

* Patients who have corneal melt, corneal epitheliopathy, abnormal corneal epithelial wound healing.
* Patients who are pregnancy or lactation.
* Patients who have a history of allergy to bevacizumab.
* Patients who have a history of allergy to steroid eye drops

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2010-12; Primary Completion 2013-03 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
rate of recurrence after primary pterygium removal | 3 months

SECONDARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | 3 months
  Local and systemic adverse events will be evaluated once a month. Number of participants with adverse events will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Ngamjit Kasetsuwan, MD, Principal Investigator — Chulalongkorn Universitiy
Locations (1):
- Faculty of medicine, Chulalongkorn university, Pathumwan, Bangkok, Thailand

REFERENCES:
- [Derived] Kasetsuwan N, Reinprayoon U, Satitpitakul V. Prevention of recurrent pterygium with topical bevacizumab 0.05% eye drops: a randomized controlled trial. Clin Ther. 2015 Oct 1;37(10):2347-51. doi: 10.1016/j.clinthera.2015.08.023. Epub 2015 Sep 26. PMID 26409291